CLINICAL TRIAL: NCT04343560
Title: Effects of Abnormal Steroid Metabolome on Bone Strength and Quality, Bone Density, Bone Remodeling, and Body Composition in Patients With MACS and Healthy Volunteers.
Brief Title: MACS and Healthy Volunteers Bone Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Irina Bancos, Principal Investigator, Mayo Clinic
Other Study IDs: 18-009787
Record Dates: First submitted 2020-04-10; First posted 2020-04-13 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: MACS Syndrome
MeSH Terms: conditions — Macrocephaly, Alopecia, Cutis Laxa, and Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 24 hour urine collection in day and night containers. Serum blood to be analyzed for PTH, sclerostin, Ca, P, CTX, osteocalcin, PINP, Total and free cortisol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with MACS: Patients with adrenal adenoma and dexamethasone suppression test >1.8 mcg/dl
- healthy controls: no history of adrenal and pituitary disease, no exogenous steroids

SUMMARY:
Adrenal adenoma is detected in 5-7% of adults and demonstrates mild autonomous cortisol secretion (MACS, dexamethasone suppression test >1.8 mcg/dl) in 50% of individuals with adenoma. Published reports suggest a 48%-52% 2-year incidence of new vertebral fractures in patients with MACS without any significant changes in bone density measurements. A disproportionate decrease in bone quality versus density or other factors such as sarcopenia potentially contribute to development of new vertebral fractures. Determining which specific abnormalities in the steroid metabolome affect bone density, quality and strength as well as bone remodeling markers and body composition will potentially serve as a diagnostic biomarker of clinical significance.

DETAILED DESCRIPTION:
In this study, we will determine whether patients with MACS (versus healthy age and sex matched controls) demonstrate: 1) decreased bone strength and quality disproportionate to the decrease of bone density and 2) abnormalities in the steroid metabolome correlate with the degree of abnormalities in bone parameters. In a cross-sectional study of 75 patients with MACS and 75 age- and sex-matched healthy controls, we will determine the relationship of the steroid metabolome to measurements of bone density, quality and strength, bone turnover markers, as well as body composition. All patients will be interviewed in regards to their health, to include questions on bone health, frailty, cognition (NIH toolbox), and quality of life. We will measure 1) BMD (bone mineral density) at the lumbar spine, hip and radius and body composition using dual-energy X ray absorptiometry (DXA), 2) radial and tibial bone microstructure by high-resolution peripheral quantitative computed tomography (HR-pQCT), 4) bone turnover markers (osteocalcin, PINP, CTx, sclerostin). 5) Age reader measurement, 6) hand grip measurement, 7) 6 minute walk test. All patients will provide a 24 h urine for steroid metabolome analysis. For primary outcomes, we will determine if steroid metabolome profiling better predicts abnormal bone strength (as measured by trabecular bone volume/tissue volume [BV/TV] ratio).

ELIGIBILITY:
Inclusion Criteria:

* Patients with MACS
* Age 18-no maximum
* exogenous steroids therapy within the last 5 years ( for more than 3 months , prednisone equivalent >7.5 mg daily)
* steroid hormone replacement therapy
* any drug therapy affecting bone metabolism
* recent fracture

Exclusion Criteria:

* exogenous steroids therapy within the last 5 years ( for more than 3 months , prednisone equivalent >7.5 mg daily)
* steroid hormone replacement therapy ( for adrenal insufficiency, hypogonadism, menopause)
* therapy for osteoporosis
* any drug therapy affecting bone metabolism
* comorbidities affecting steroid metabolome or bone metabolism
* recent fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MACS participants either male or female who are at least 18 years of age who fulfill the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
BV/TV ratio | 0-24 months
  measured by computed tomography
steroid metabolome | 0-24 months
  24h urine steroid profiling

CONTACTS AND LOCATIONS:
Overall Officials: Irina Bancos, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials